CLINICAL TRIAL: NCT01096667
Title: A 4-Week, Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Parallel Group Study To Evaluate The Safety, Tolerability And Efficacy Of Once Daily PF-04971729 And Hydrochlorothiazide In Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic And Blood Pressure Control
Brief Title: Study of Safety and Efficacy Of Ertugliflozin (PF-04971729, MK-8835) In Participants With Type 2 Diabetes And Hypertension (MK-8835-042)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8835-042; B1521004 (Other: Pfizer protocol number); MK-8835-042 (Other: Merck Protocol Number)
Record Dates: First submitted 2010-03-26; First posted 2010-03-31 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
Keywords: type 2 diabetes; hypertension; ambulatory blood pressure monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — ertugliflozin; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo to ertugliflozin (resembling either 1 mg or 5 mg), placebo to ertugliflozin (resembling 25 mg), and placebo to HCTZ once daily for 28 days.
  Interventions: Drug: Placebo to Ertuglilflozin 1 or 5 mg; Drug: Placebo to HCTZ; Drug: Placebo to ertuglilflozin 25 mg
- Ertugliflozin 1 mg (Experimental): Ertugliflozin 1 mg, placebo to ertugliflozin (resembling 25 mg), and placebo to HCTZ once daily for 28 days
  Interventions: Drug: Ertugliflozin 1 mg; Drug: Placebo to HCTZ; Drug: Placebo to ertuglilflozin 25 mg
- Ertugliflozin 5 mg (Experimental): Ertugliflozin 5 mg, placebo to ertugliflozin (resembling 25 mg), and placebo to HCTZ once daily for 28 days
  Interventions: Drug: Ertugliflozin 5 mg; Drug: Placebo to HCTZ; Drug: Placebo to ertuglilflozin 25 mg
- Ertugliflozin 25 mg (Experimental): Ertugliflozin 25 mg, placebo to ertugliflozin (resembling either 1 mg or 5 mg), and placebo to HCTZ once daily for 28 days
  Interventions: Drug: Placebo to Ertuglilflozin 1 or 5 mg; Drug: Ertugliflozin 25 mg; Drug: Placebo to HCTZ
- HCTZ 12.5mg (Active Comparator): HCTZ 12.5 mg, placebo to ertugliflozin (resembling either 1 mg or 5 mg), and placebo to ertugliflozin (resembling 25 mg) once daily for 28 days
  Interventions: Drug: Placebo to Ertuglilflozin 1 or 5 mg; Drug: HCTZ 12.5mg; Drug: Placebo to ertuglilflozin 25 mg

INTERVENTIONS:
Drug: Placebo to Ertuglilflozin 1 or 5 mg — Placebo to ertuglilflozin tablet 1 or 5 mg once daily for 28 days
  Arms: Ertugliflozin 25 mg; HCTZ 12.5mg; Placebo
Drug: Ertugliflozin 1 mg — Ertugliflozin tablet 1 mg once daily for 28 days
  Arms: Ertugliflozin 1 mg
Drug: Ertugliflozin 5 mg — Ertugliflozin tablet 5 mg once daily for 28 days
  Arms: Ertugliflozin 5 mg
Drug: Ertugliflozin 25 mg — Ertugliflozin tablet 25 mg once daily for 28 days
  Arms: Ertugliflozin 25 mg
Drug: HCTZ 12.5mg — Hydrocholorthiazide (HCTZ) 12.5 mg capsule once daily for 28 days
  Arms: HCTZ 12.5mg
Drug: Placebo to HCTZ — Placebo to HCTZ 12.5 mg capsule once daily for 28 days
  Arms: Ertugliflozin 1 mg; Ertugliflozin 25 mg; Ertugliflozin 5 mg; Placebo
Drug: Placebo to ertuglilflozin 25 mg — Placebo to ertuglilflozin tablet 25 mg once daily for 28 days
  Arms: Ertugliflozin 1 mg; Ertugliflozin 5 mg; HCTZ 12.5mg; Placebo

SUMMARY:
MK-8835-042 (B1521004) is designed to assess the safety and efficacy of an investigational drug, ertugliflozin (MK-8835, PF-04971729), in participants with type 2 diabetes and hypertension. Participants in the study will receive 1 of 5 treatments for 28 days (either placebo, 1 of 3 doses of ertugliflozin [1, 5, or 25 mg], or the approved drug hydrochlorothiazide [HCTZ]). The primary hypothesis of the study was that ertugliflozin was superior to placebo on the change from baseline in average, 24-hour systolic blood pressure (SBP) on Day 28.

ELIGIBILITY:
Inclusion Criteria:

* Participants with type 2 diabetes and hypertension
* Medically stable
* On at least 1 (and up to 2) oral diabetes drugs
* And up to 2 medicines for blood pressure control

Exclusion Criteria:

* Participants with type 1 diabetes
* Heart attack
* Stroke
* Uncontrolled blood pressure
* Significant kidney disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2010-05-17 (Actual); Primary Completion 2011-02-09 (Actual); Study Completion 2011-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Amin NB, Wang X, Mitchell JR, Lee DS, Nucci G, Rusnak JM. Blood pressure-lowering effect of the sodium glucose co-transporter-2 inhibitor ertugliflozin, assessed via ambulatory blood pressure monitoring in patients with type 2 diabetes and hypertension. Diabetes Obes Metab. 2015 Aug;17(8):805-8. doi: 10.1111/dom.12486. Epub 2015 Jun 17. PMID 25951755
- [Derived] Fediuk DJ, Sahasrabudhe V, Dawra VK, Zhou S, Sweeney K. Population Pharmacokinetic Analyses of Ertugliflozin in Select Ethnic Populations. Clin Pharmacol Drug Dev. 2021 Nov;10(11):1297-1306. doi: 10.1002/cpdd.970. Epub 2021 Jul 2. PMID 34213819

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, 194 participants received placebo for at least 3 weeks (completed the run-in period). Treated participants included all randomized participants who received at least one dose of study drug.
Groups:
- Placebo: Placebo for Ertugliflozin (1 mg or 5 mg and 25 mg) and placebo to hydrochlorothiazide (HCTZ), once daily for 28 days.
- Ertugliflozin 1 mg: Ertugliflozin 1 mg, placebo to ertugliflozin (25 mg), and placebo to HCTZ, once daily for 28 days
- Ertugliflozin 5 mg: Ertugliflozin 5 mg, placebo to ertugliflozin (25 mg), and placebo to HCTZ, once daily for 28 days
- Ertugliflozin 25 mg: Ertugliflozin 25 mg, placebo to ertugliflozin (1 mg or 5 mg), and placebo to HCTZ, once daily for 28 days
- HCTZ 12.5mg: HCTZ 12.5 mg, placebo to ertugliflozin (1 mg or 5 mg and 25 mg), once daily for 28 days
Period: Overall Study
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Started | 39 | 39 | 38 | 39 | 39
Treated | 38 | 39 | 38 | 39 | 39
Completed | 36 | 37 | 36 | 36 | 39
Not Completed | 3 | 2 | 2 | 3 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0
Not completed — Reason not available | 0 | 1 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Not treated | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population includes participants who received at least 1 dose of blinded treatment regimen.
Groups:
- Placebo: Placebo for Ertugliflozin (1 mg or 5 mg and 25 mg) and placebo to HCTZ, once daily for 28 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg | Total
Number analyzed (Participants) | 38 | 39 | 38 | 39 | 39 | 193
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 44 years | 3 | 4 | 3 | 5 | 1 | 16
  Between 45 and 64 years | 34 | 34 | 32 | 34 | 34 | 168
  65 years and older | 1 | 1 | 3 | 0 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 13 | 12 | 11 | 62
  Male | 24 | 27 | 25 | 27 | 28 | 131

OUTCOME MEASURES:

1. Primary Outcome: Baseline 24-hour Average Systolic Blood Pressure (SBP)
Description: Baseline 24-hour average SBP was assessed using 24-hour ambulatory blood pressure monitoring (ABPM).
Time Frame: 24 hours
Population: All randomized participants who received at least one dose of study drug and had a baseline measurement for average 24-hour SBP.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 37 | 39 | 38 | 39 | 38
mmHg | 136.11 (15.298) | 133.13 (10.868) | 135.08 (12.073) | 135.59 (11.929) | 139.55 (11.941)

2. Primary Outcome: Change From Baseline on 24-hour Average SBP at Week 4
Description: Change from baseline on 24-hour average SBP at Week 4 assessed using 24-hour ABPM. In the case of missing data, last observation carried forward (LOCF).
Time Frame: Baseline and Week 4
Population: Analysis population consisted of all randomized participants who received at least 1 dose of blinded treatment and had baseline measurement and a post-randomization measurement for average, 24-hour SBP.
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 30 | 35 | 28 | 33 | 34
mmHg | 0.26 [-1.31 to 1.70] | -2.71 [-4.15 to -1.33] | -3.73 [-5.30 to -2.18] | -3.42 [-4.86 to -1.99] | -2.95 [-4.39 to -1.51]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.034, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -2.97, 80% CI 2-sided [-5.05 to -0.89]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.010, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -4.00, 80% CI 2-sided [-6.17 to -1.82]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.012, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -3.69, 80% CI 2-sided [-5.78 to -1.60]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.024, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -3.21, 80% CI 2-sided [-5.30 to -1.13]

3. Secondary Outcome: Baseline Average Daytime and Nighttime SBP
Description: Daytime was defined as 0600 to 2159 hours, inclusive, local time. Nighttime was defined as 2200 to 0559 hours, inclusive, local time.
Time Frame: Daytime: 16 hours; Nighttime: 8 hours
Population: All randomized participants who received at least one dose of study drug and had a baseline measurement for daytime and nighttime SBP.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 37 | 39 | 38 | 39 | 38
mmHg
  Daytime | 139.95 (15.107) | 136.85 (11.361) | 138.89 (11.724) | 139.56 (12.343) | 143.32 (12.637)
  Nighttime | 127.54 (16.858) | 125.15 (12.180) | 126.37 (13.956) | 127.13 (13.553) | 131.68 (12.912)

4. Secondary Outcome: Change From Baseline on Daytime Average SBP at Week 4
Description: Change from baseline on daytime average SBP at Week 4 using 24 hour ABPM. In the case of missing data, LOCF. Daytime was defined as 0600 to 2159 hours, inclusive, local time.
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 30 | 35 | 28 | 33 | 34
mmHg | 0.82 [-0.90 to 2.34] | -2.88 [-4.49 to -1.44] | -3.61 [-5.30 to -1.94] | -4.17 [-5.72 to -2.63] | -3.10 [-4.66 to -1.57]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.018, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -3.70, 80% CI 2-sided [-5.94 to -1.46]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.008, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -4.43, 80% CI 2-sided [-6.78 to -2.09]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -4.99, 80% CI 2-sided [-7.24 to -2.74]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.013, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -3.92, 80% CI 2-sided [-6.16 to -1.67]

5. Secondary Outcome: Change From Baseline on Nighttime Average SBP at Week 4
Description: Change from baseline on nighttime average SBP at Week 4 using 24 hour ABPM. In the case of missing data, LOCF. Nighttime was defined as 2200 to 0559 hours, inclusive, local time.
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 30 | 35 | 28 | 33 | 34
mmHg | -0.29 [-2.28 to 1.71] | -2.48 [-4.33 to -0.60] | -3.47 [-5.53 to -1.39] | -2.31 [-4.21 to -0.40] | -2.30 [-4.20 to -0.40]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.152, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -2.19, 80% CI 2-sided [-4.93 to 0.54]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.078, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -3.18, 80% CI 2-sided [-6.06 to -0.30]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.174, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -2.02, 80% CI 2-sided [-4.79 to 0.74]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.174, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -2.01, 80% CI 2-sided [-4.77 to 0.74]

6. Secondary Outcome: Baseline Seated, Triplicate Trough SBP
Description: Trough SBP was measured using an automated blood pressure device with the participant in a seated position for at least 5 minutes before and while the blood pressure measure is obtained. Three measurements of blood pressure were taken at least 2-minutes apart. Baseline trough SBP is calculated as the mean of triplicate (3) trough SBP measures.
Time Frame: Baseline
Population: All randomized participants who received at least one dose of study drug and had a baseline measurement for seated, triplicate, trough SBP.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 38 | 39 | 38 | 39 | 39
mmHg | 135.17 (14.183) | 134.23 (13.631) | 137.31 (14.834) | 135.25 (13.452) | 138.07 (12.958)

7. Secondary Outcome: Change From Baseline in Seated, Triplicate Trough SBP at Week 4
Description: Trough SBP was measured using an automated blood pressure device with the participant in a seated position for at least 5 minutes before and while the blood pressure measure is obtained. Three measurements of blood pressure were taken at least 2-minutes apart. The change from baseline at Week 4 is the difference between the baseline and Week 4 assessments.
Time Frame: Baseline and Week 4
Population: Analysis population consisted of all randomized participants who received at least 1 dose of blinded treatment and had baseline measurement and post-randomization measurement for sitting, triplicate trough SBP.
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 37 | 37 | 36 | 36 | 39
mmHg | 1.24 [-0.93 to 3.41] | -2.77 [-4.95 to -0.60] | -5.92 [-8.12 to -3.73] | -4.96 [-7.15 to -2.77] | -3.13 [-5.26 to -1.00]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.047, Mixed Model for Repeated Measures — P-value is one-sided; With terms for treatment, visit, and treatment-by-visit interaction as fixed effects, participant as random effect and baseline as the covariate; Difference in least squares means = -4.01, 80% CI 2-sided [-7.09 to -0.94]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.002, Mixed Model for Repeated Measures — P-value is one-sided; [statistical method as in outcome 7, analysis 1]; Difference in least squares means = -7.16, 80% CI 2-sided [-10.25 to -4.07]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.005, Mixed Model for Repeated Measures — P-value is one-sided; [statistical method as in outcome 7, analysis 1]; Difference in least squares means = -6.20, 80% CI 2-sided [-9.28 to -3.11]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.033, Mixed Model for Repeated Measures — P-value is one-sided; [statistical method as in outcome 7, analysis 1]; Difference in least squares means = -4.37, 80% CI 2-sided [-7.41 to -1.33]

8. Secondary Outcome: Baseline 24-hour, Daytime and Nightime Average Diastolic Blood Pressure (DBP)
Description: Baseline 24-hour average DBP was assessed using 24-hour ABPM. Daytime was defined as 0600 to 2159 hours, inclusive, local time. Nighttime was defined as 2200 to 0559 hours, inclusive, local time.
Time Frame: up to 24 hours
Population: All randomized participants who received at least one dose of study drug and had a baseline measurement for average 24-hour, daytime and nighttime DBP.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 37 | 39 | 38 | 39 | 38
mmHg
  24-hr | 81.89 (9.655) | 78.67 (8.600) | 80.18 (8.655) | 80.36 (8.650) | 82.66 (9.459)
  Daytime | 85.32 (10.127) | 81.77 (8.925) | 83.47 (9.164) | 83.59 (9.295) | 85.87 (9.884)
  Nighttime | 74.24 (9.717) | 72.05 (9.330) | 73.05 (9.034) | 73.28 (8.760) | 75.76 (10.042)

9. Secondary Outcome: Change From Baseline on 24-hour Average DBP at Week 4
Description: Change from baseline on 24-hour average DBP at Week 4 using 24 hour ABPM. In the case of missing data, LOCF.
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 30 | 35 | 28 | 33 | 34
mmHg | 0.77 [-0.25 to 1.75] | -1.89 [-2.81 to -0.95] | -2.34 [-3.37 to -1.31] | -1.50 [-2.45 to -0.55] | -1.42 [-2.37 to -0.48]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.007, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate. p-value is one-sided; Difference in least squares means = -2.66, 80% CI 2-sided [-4.03 to -1.29]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate. p-value is one-sided; Difference in least squares means = -3.11, 80% CI 2-sided [-4.55 to -1.67]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.018, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate. p-value is one-sided; Difference in least squares means = -2.27, 80% CI 2-sided [-3.65 to -0.88]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.021, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate. p-value is one-sided; Difference in least squares means = -2.19, 80% CI 2-sided [-3.56 to -0.82]

10. Secondary Outcome: Change From Baseline on Daytime Average DBP at Week 4
Description: Change from baseline on daytime average DBP at Week 4 using 24 hour ABPM. In the case of missing data, LOCF. Daytime was defined as 0600 to 2159 hours, inclusive, local time.
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 30 | 35 | 28 | 33 | 34
mmHg | 0.87 [-0.24 to 1.85] | -2.12 [-3.13 to -1.18] | -1.88 [-2.96 to -0.80] | -1.77 [-2.77 to -0.78] | -1.69 [-2.67 to -0.70]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate. p-value is one-sided; Difference in least squares means = -2.99, 80% CI 2-sided [-4.43 to -1.55]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.010, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate. p-value is one-sided; Difference in least squares means = -2.75, 80% CI 2-sided [-4.26 to -1.24]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.010, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate. p-value is one-sided; Difference in least squares means = -2.64, 80% CI 2-sided [-4.09 to -1.19]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.011, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate. p-value is one-sided; Difference in least squares means = -2.57, 80% CI 2-sided [-4.00 to -1.13]

11. Secondary Outcome: Change From Baseline on Nighttime Average DBP at Week 4
Description: Change from baseline on nighttime average DBP at Week 4 using 24 hour ABPM. In the case of missing data, LOCF. Nighttime was defined as 2200 to 0559 hours, inclusive, local time.
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 30 | 35 | 28 | 33 | 34
mmHg | 1.02 [-0.39 to 2.44] | -1.48 [-2.78 to -0.15] | -2.52 [-3.98 to -1.06] | -0.84 [-2.19 to 0.51] | -0.55 [-1.95 to 0.71]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.048, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -2.50, 80% CI 2-sided [-4.43 to -0.57]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.013, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -3.54, 80% CI 2-sided [-5.58 to -1.51]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.111, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -1.88, 80% CI 2-sided [-3.82 to 0.09]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.148, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -1.58, 80% CI 2-sided [-3.51 to 0.36]

12. Secondary Outcome: Baseline Seated, Triplicate Trough DBP
Description: Trough DBP was measured using an automated blood pressure device with the participant in a seated position for at least 5 minutes before and while the blood pressure measure is obtained. Three measurements of blood pressure were taken at least 2-minutes apart. Baseline trough DBP is calculated as the mean of triplicate (3) trough DBP measures.
Time Frame: Baseline
Population: All randomized participants who received at least one dose of study drug and had a baseline measurement for seated, triplicate, trough DBP.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 38 | 39 | 38 | 39 | 39
mmHg | 84.89 (9.462) | 83.08 (7.557) | 83.79 (7.904) | 83.89 (8.290) | 84.72 (8.043)

13. Secondary Outcome: Change From Baseline in Seated, Triplicate Trough DBP at Week 4
Description: Trough DBP was measured using an automated blood pressure device with the participant in a seated position for at least 5 minutes before and while the blood pressure measure is obtained. Three measurements of blood pressure were taken at least 2-minutes apart. The change from baseline at Week 4 is the difference between the baseline and Week 4 assessments.
Time Frame: Baseline and Week 4
Population: Analysis population consisted of all randomized participants who received at least 1 dose of blinded treatment and had baseline measurement and post-randomization measurement for sitting, triplicate trough DBP.
Measure: Least Squares Mean (80% Confidence Interval); unit: mmHg
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 37 | 37 | 36 | 36 | 39
mmHg | 0.30 [-0.97 to 1.58] | -0.90 [-2.18 to 0.37] | -0.75 [-2.03 to 0.54] | -2.71 [-4.00 to -1.43] | -2.54 [-3.79 to -1.29]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.196, Mixed Measures Repeated Model — P-value is one-sided; [statistical method as in outcome 7, analysis 1]; Difference in least squares means = -1.20, 80% CI 2-sided [-3.01 to 0.60]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.229, Mixed Measures Repeated Model — P-value is one-sided; [statistical method as in outcome 7, analysis 1]; Difference in least squares means = -1.05, 80% CI 2-sided [-2.86 to 0.77]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.017, Mixed Measures Repeated Model — P-value is one-sided; [statistical method as in outcome 7, analysis 1]; Difference in least squares means = -3.02, 80% CI 2-sided [-4.83 to -1.20]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.021, Mixed Measures Repeated Model — P-value is one-sided; [statistical method as in outcome 7, analysis 1]; Difference in least squares means = -2.84, 80% CI 2-sided [-4.63 to -1.06]

14. Secondary Outcome: Baseline 24-hour, Daytime and Nightime Average Heart Rate
Description: Baseline 24-hour average heart rate was assessed using 24-hour ABPM. Daytime was defined as 0600 to 2159 hours, inclusive, local time. Nighttime was defined as 2200 to 0559 hours, inclusive, local time.
Time Frame: up to 24 hours
Population: All randomized participants who received at least one dose of study drug and had a baseline measurement for average 24-hour, daytime and nighttime heart rate.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 37 | 39 | 38 | 39 | 38
beats per minute
  24-hr | 81.11 (9.486) | 80.74 (6.950) | 79.68 (10.081) | 79.41 (9.063) | 79.08 (9.216)
  Daytime | 84.43 (9.743) | 83.74 (7.044) | 82.71 (10.405) | 82.18 (9.136) | 81.95 (9.470)
  Nighttime | 74.05 (9.871) | 74.44 (8.133) | 73.16 (10.205) | 73.49 (10.034) | 73.03 (9.736)

15. Secondary Outcome: Change From Baseline on 24-hour Average Heart Rate at Week 4
Description: Change from baseline in 24-hour average heart rate at Week 4 using 24 hour ABPM.
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Least Squares Mean (80% Confidence Interval); unit: Beats per minute
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 30 | 35 | 28 | 33 | 34
Beats per minute | 1.00 [-0.21 to 2.16] | -1.22 [-2.45 to -0.25] | 1.07 [-0.16 to 2.29] | -1.39 [-2.52 to -0.26] | -0.56 [-1.68 to 0.56]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.039, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -2.22, 80% CI 2-sided [-3.83 to -0.61]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.521, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = 0.07, 80% CI 2-sided [-1.63 to 1.77]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.031, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -2.39, 80% CI 2-sided [-4.02 to -0.75]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.110, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -1.56, 80% CI 2-sided [-3.19 to 0.07]

16. Secondary Outcome: Change From Baseline on Daytime Average Heart Rate at Week 4
Description: Change from baseline in daytime average heart rate at Week 4 using 24 hour ABPM. In the case of missing data, LOCF. Daytime was defined as 0600 to 2159 hours, inclusive, local time.
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Least Squares Mean (80% Confidence Interval); unit: Beats per minute
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 30 | 35 | 28 | 33 | 34
Beats per minute | 1.58 [0.25 to 2.83] | -1.80 [-3.09 to -0.70] | 1.10 [-0.24 to 2.43] | -1.07 [-2.31 to 0.15] | -0.06 [-1.22 to 1.22]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.007, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -3.38, 80% CI 2-sided [-5.13 to -1.63]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.370, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -0.48, 80% CI 2-sided [-2.33 to 1.38]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.029, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -2.65, 80% CI 2-sided [-4.43 to -0.87]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.118, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -1.64, 80% CI 2-sided [-3.42 to 0.13]

17. Secondary Outcome: Change From Baseline on Nighttime Average Heart Rate at Week 4
Description: Change from baseline in 24-hour nighttime average heart rate at Week 4 using 24 hour ABPM. In the case of missing data, LOCF. Nighttime was defined as 2200 to 0559 hours, inclusive, local time.
Time Frame: Baseline and Week 4
Population: as for outcome 2
Measure: Least Squares Mean (80% Confidence Interval); unit: Beats per minute
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 30 | 35 | 28 | 33 | 34
Beats per minute | -0.18 [-1.63 to 1.25] | -0.15 [-1.76 to 0.91] | 1.43 [-0.07 to 2.92] | -1.99 [-3.38 to -0.63] | -1.24 [-2.70 to 0.00]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.506, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = 0.02, 80% CI 2-sided [-1.96 to 2.00]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.838, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = 1.61, 80% CI 2-sided [-0.49 to 3.71]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.123, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -1.82, 80% CI 2-sided [-3.82 to 0.19]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.246, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -1.07, 80% CI 2-sided [-3.06 to 0.93]

18. Secondary Outcome: Baseline Seated, Triplicate Trough Heart Rate
Description: Trough heart rate was measured using an automated blood pressure device with the participant in a seated position for at least 5 minutes before and while the heart rate measure was obtained. Three measurements of heart rate were taken at least 2-minutes apart. Baseline trough heart rate is calculated as the mean of triplicate (3) trough heart rate measures.
Time Frame: Baseline
Population: All randomized participants who received at least one dose of study drug and had a baseline measurement for seated, triplicate, trough heart rate.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 38 | 39 | 38 | 39 | 39
beats per minute | 77.07 (9.713) | 78.73 (8.446) | 77.30 (11.749) | 75.63 (9.550) | 77.97 (11.462)

19. Secondary Outcome: Change From Baseline in Seated, Triplicate Trough Heart Rate at Week 4
Description: Trough heart rate was measured using an automated blood pressure device with the participant in a seated position for at least 5 minutes before and while the heart rate measure was obtained. Three measurements of heart rate were taken at least 2-minutes apart. The change from baseline at Week 4 is the difference between the baseline and Week 4 assessments.
Time Frame: Baseline and Week 4
Population: Analysis population consisted of all randomized participants who received at least 1 dose of blinded treatment and had baseline measurement and post-randomization measurement for sitting, triplicate trough heart rate.
Measure: Least Squares Mean (80% Confidence Interval); unit: beats per minute
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 37 | 37 | 36 | 36 | 39
beats per minute | 2.34 [0.85 to 3.82] | -1.86 [-3.35 to -0.38] | 1.22 [-0.28 to 2.71] | -1.51 [-3.01 to -0.01] | -0.99 [-2.44 to 0.46]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.005, Mixed Model for Repeated Measures — P-value is one-sided; [statistical method as in outcome 7, analysis 1]; Difference in least squares means = -4.20, 80% CI 2-sided [-6.30 to -2.10]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.248, Mixed Model for Repeated Measures — P-value is one-sided; [statistical method as in outcome 7, analysis 1]; Difference in least squares means = -1.12, 80% CI 2-sided [-3.23 to 0.99]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.010, Mixed Model for Repeated Measures — P-value is one-sided; [statistical method as in outcome 7, analysis 1]; Difference in least squares means = -3.84, 80% CI 2-sided [-5.95 to -1.73]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.020, Mixed Model for Repeated Measures — P-value is one-sided; [statistical method as in outcome 7, analysis 1]; Difference in least squares means = -3.33, 80% CI 2-sided [-5.40 to -1.25]

20. Secondary Outcome: Baseline 24-hour Average Urinary Glucose Excretion
Description: Urinary glucose excetion was corrected for a duration of 24 hours (with appropriate duration of collection defined as >20 hours and <28 hours).
Time Frame: 24 hours
Population: All randomized participants who received at least one dose of study drug and had a baseline measurement for average urinary glucose excretion
Measure: Mean (Standard Deviation); unit: grams/day
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 36 | 38 | 37 | 39 | 39
grams/day | 13.35 (22.913) | 9.97 (20.085) | 8.04 (13.135) | 17.56 (29.101) | 6.96 (8.562)

21. Secondary Outcome: Change From Baseline on 24-hour Urinary Glucose Excretion at Week 4
Description: Urinary glucose excetion was corrected for a duration of 24 hours (with appropriate duration of collection defined as >20 hours and <28 hours). In the case of missing data, LOCF.
Time Frame: Baseline and Week 4
Population: Analysis population consisted of all randomized participants who received at least 1 dose of blinded treatment and had baseline measurement and post-randomization measurement for 24-hour urinary glucose excretion.
Measure: Least Squares Mean (80% Confidence Interval); unit: grams/day
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 35 | 36 | 34 | 36 | 39
grams/day | 4.15 [-3.50 to 11.81] | 46.33 [38.79 to 53.88] | 64.54 [56.77 to 72.31] | 74.49 [66.87 to 82.11] | -0.48 [-7.76 to 6.80]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value rounded to thousandths; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = 42.18, 80% CI 2-sided [31.42 to 52.94]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value rounded to thousandths; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = 60.39, 80% CI 2-sided [49.47 to 71.31]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.000, ANCOVA — P-value is one-sided. P-value rounded to thousandths; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = 70.34, 80% CI 2-sided [59.58 to 81.10]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.713, ANCOVA — P-value is one-sided; Based on ANCOVA with treatment as fixed effect and baseline as a covariate; Difference in least squares means = -4.63, 80% CI 2-sided [-15.22 to 5.96]

22. Secondary Outcome: Baseline Fasting Plasma Glucose (FPG)
Description: For FPG, blood was drawn after an overnight fast of at least 8 hours (except water).
Time Frame: Baseline
Population: All randomized participants.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 38 | 39 | 38 | 39 | 39
mg/dL | 169.47 (51.073) | 158.38 (40.806) | 158.29 (42.465) | 172.03 (55.878) | 156.87 (36.541)

23. Secondary Outcome: Change From Baseline in FPG at Week 4
Description: For FPG, blood was drawn after an overnight fast of at least 8 hours (except water).
Time Frame: Baseline and Week 4
Population: Analysis population consisted of all randomized participants who received at least 1 dose of blinded treatment and had baseline measurement and post-randomization measurement at Week 4 for FPG (observed cases).
Measure: Least Squares Mean (80% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 37 | 36 | 35 | 35 | 37
mg/dL | 4.39 [-2.16 to 10.94] | -13.70 [-20.35 to -7.06] | -30.41 [-37.12 to -23.71] | -31.03 [-37.74 to -24.32] | 3.79 [-2.74 to 10.31]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.007, Mixed Model for Repeated Measures — P-value is one-sided; With treatment, visit, and treatment-by-visit interaction as fixed effects, participant as random effect and baseline FPG as the covariate; Difference in least squares means = -18.10, 80% CI 2-sided [-27.45 to -8.75]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.000, Mixed Model for Repeated Measures — P-value is one-sided. P-value rounded to thousandths; [statistical method as in outcome 23, analysis 1]; Difference in least squares means = -34.81, 80% CI 2-sided [-44.19 to -25.43]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.000, Mixed Model for Repeated Measures — P-value is one-sided. P-value rounded to thousandths; [statistical method as in outcome 23, analysis 1]; Difference in least squares means = -35.42, 80% CI 2-sided [-44.78 to -26.07]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.467, Mixed Model for Repeated Measures — P-value is one-sided; [statistical method as in outcome 23, analysis 1]; Difference in least squares means = -0.61, 80% CI 2-sided [-9.86 to 8.65]

24. Secondary Outcome: Change From Baseline in FPG at Week 2
Description: For FPG, blood was drawn after an overnight fast of at least 8 hours (except water).
Time Frame: Baseline and Week 2
Population: Analysis population consisted of all randomized participants who received at least 1 dose of blinded treatment and had baseline measurement and post-randomization measurement at Week 2 for FPG (observed cases).
Measure: Least Squares Mean (80% Confidence Interval); unit: mg/dL
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 38 | 35 | 34 | 36 | 37
mg/dL | -5.44 [-11.93 to 1.04] | -10.98 [-17.69 to -4.26] | -22.45 [-29.23 to -15.67] | -32.03 [-38.66 to -25.40] | 3.21 [-3.32 to 9.74]
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin 1 mg; Test type: Superiority or Other; p = 0.224, Mixed Model for Repeated Measures — P-value is one-sided; [statistical method as in outcome 23, analysis 1]; Difference in least squares means = -5.54, 80% CI 2-sided [-14.89 to 3.82]
Statistical Analysis 2: Comparison: Placebo vs Ertugliflozin 5 mg; Test type: Superiority or Other; p = 0.011, Mixed Model for Repeated Measures — P-value is one-sided; [statistical method as in outcome 23, analysis 1]; Difference in least squares means = -17.00, 80% CI 2-sided [-26.39 to -7.61]
Statistical Analysis 3: Comparison: Placebo vs Ertugliflozin 25 mg; Test type: Superiority or Other; p = 0.000, Mixed Model for Repeated Measures — P-value is one-sided. P-value rounded to thousandths; [statistical method as in outcome 23, analysis 1]; Difference in least squares means = -26.59, 80% CI 2-sided [-35.84 to -17.33]
Statistical Analysis 4: Comparison: Placebo vs HCTZ 12.5mg; Test type: Superiority or Other; p = 0.886, Mixed Model for Repeated Measures — P-value is one-sided; [statistical method as in outcome 23, analysis 1]; Difference in least squares means = 8.65, 80% CI 2-sided [-0.56 to 17.87]

25. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. The table below includes all data collected since first dose of study drug.
Time Frame: Up to 63 days (including run-in, treatment period, and follow-up)
Population: Analysis population consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 38 | 39 | 38 | 39 | 39
Participants | 9 | 8 | 15 | 12 | 10

26. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An adverse event is defined as any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. The table below includes all data collected since first dose of study drug. Discontinuation of study drug due to an AE includes temporary and permanent discontinuation of study drug due to an AE.
Time Frame: Up to 28 days (treatment period)
Population: Analysis population consisted of all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg
Number analyzed (Participants) | 38 | 39 | 38 | 39 | 39
Participants | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 63 days (including screening and run-in [pre-randomization], treatment period, and follow-up)
Description: Serious adverse events include all randomized participants who received at least one dose of study drug except for the pre-randomization arm that includes all randomized participants. Non-serious adverse events include all randomized participants who received at least one dose of study drug (all arms).
Groups:
- Pre-randomization: Blinded placebo was administered for at least 21 days prior to randomization.
Arm/Group | Placebo | Ertugliflozin 1 mg | Ertugliflozin 5 mg | Ertugliflozin 25 mg | HCTZ 12.5mg | Pre-randomization
Serious Adverse Events (participants affected / at risk) | 1/38 | 0/39 | 0/38 | 0/39 | 0/39 | 1/194
Other Adverse Events (participants affected / at risk) | 3/38 | 4/39 | 8/38 | 6/39 | 6/39 | 10/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=38) | Ertugliflozin 1 mg (N=39) | Ertugliflozin 5 mg (N=38) | Ertugliflozin 25 mg (N=39) | HCTZ 12.5mg (N=39) | Pre-randomization (N=194)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=38) | Ertugliflozin 1 mg (N=39) | Ertugliflozin 5 mg (N=38) | Ertugliflozin 25 mg (N=39) | HCTZ 12.5mg (N=39) | Pre-randomization (N=193)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Athralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator will provide manuscripts, abstracts, or the full text of any other intended disclosure (poster presentation, invited speaker or guest lecturer presentation, etc.) to the sponsor at least 30 days before they are submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, Investigator agrees to delay the disclosure for a period not to exceed an additional 60 days.